CLINICAL TRIAL: NCT06545305
Title: Incidence and Risk Factors of Ocular Complications Among Patients With Homocystinuria in Jeddah, Saudi Arabia: A Cross-sectional Study
Brief Title: Incidence and Risk Factors of Ocular Complications Among Patients With Homocystinuria
Status: Enrolling by invitation | Type: Observational
Sponsor: King Fahad Armed Forces Hospital (Other Government)
Responsible Party: Principal Investigator, Hassan A. Ahmed, Residence, King Fahad Armed Forces Hospital
Other Study IDs: Optha; King Fahd Armed Forces (Other: REC 607)
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Complications
Keywords: ocular complications; high myopia; Saudi Arabia; Classic Homocystinuria; Ectopia lentis
MeSH Terms: conditions — Homocystinuria; Ectopia Lentis | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Homocystinuria: Homocystinuria patients with Ocular complications
  Interventions: Procedure: Lensectomy and vitrectomy

INTERVENTIONS:
Procedure: Lensectomy and vitrectomy — Corrections
  Other Names: Scleral fixation; Grice green procedure

SUMMARY:
Background: Cysteine beta-synthase (CBS) deficiency, often known as classic homocystinuria (HCU), is an uncommon inborn mistake in methionine metabolism. Developmental delay, intellectual incapacity, skeletal and vascular symptoms, and ocular abnormalities are possible main clinical characteristics.

Objective: This study sought to describe the ocular anomalies that King Fahad Armed Forces Hospital, Jeddah, Saudi Arabia, HCU patients presented with between 2018 and 2022.

DETAILED DESCRIPTION:
This retrospective research included 6 HCU patients. Demographic and clinical characteristics of patients as age, gender, comorbidities were collected. Relevant clinical and ophthalmic assessments, like visual acuity, fundus examination findings, complications and type of surgery were also reported

ELIGIBILITY:
Inclusion Criteria:

* All patients from all age groups who were diagnosed with homocystinuria between 2018 and 2022 were included, regardless of whether the diagnosis was made biochemically (by exhibiting hyperhomocysteinaemia and hypermethioninaemia) or genetically (by discovering biallelic pathogenic mutations in the CBS gene)

Exclusion Criteria:

* Patients with incomplete investigations for various reasons

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patient's records gathered from outpatient internal medicine and pediatric encounters. Six patients met study inclusion criteria. Demographic and clinical characteristics of patients were collected. Relevant clinical and ophthalmic assessments, as visual acuity, fundus examination, complications and surgery type were also obtained. Visual acuity, in-clinic dilated fundus examination, optical coherence tomography (OCT) angiography, macular OCT scan, and fundus photography were components of ophthalmic examinations. Fundus examination involved retinal inspection, visual acuity measured using tumbling E chart.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Autoref reading | After one year
  Refractory errors

CONTACTS AND LOCATIONS:
Overall Officials: Hassan A Ahmed, MS, Principal Investigator — Pediatric Department, King Salman Medical city-Maternity and Children, Medina, Saudi Arabia
Locations (1):
- King Fahad Armed Forces Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The data available with principal investigator when needed